CLINICAL TRIAL: NCT05554549
Title: Risk of Hip Fracture in Meat-eaters, Pescatarians, and Vegetarians in the UK Biobank
Brief Title: Dietary Patterns and Hip Fracture Risk in the UK Biobank
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Darren Greenwood, Senior Lecturer in Biostatistics, University of Leeds
Other Study IDs: 88995
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Hip Fractures
Keywords: Nutrition; Vegetarian; Fracture; Cohort study; Epidemiology; Osteoporosis
MeSH Terms: conditions — Hip Fractures; Fractures, Bone; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — UK Biobank collected biomarker samples with DNA. This project makes use of data from the biomarker samples, but no additional samples will be taken and no additional samples will taken for this research. No samples will be processed, stored or retained by us. For the previously published details of UK Biobank, with anonymised data made available for researchers, please see: https://www.ukbiobank.ac.uk/enable-your-research/about-our-data/biomarker-data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UK Biobank: UK Biobank. There are no interventions in this observational cohort study.
  Interventions: Other: Dietary pattern observed

INTERVENTIONS:
Other: Dietary pattern observed — Dietary pattern: regular meat-eater, occasional meat-eater, pescatarian, and vegetarian. There are no interventions in this observational cohort.

SUMMARY:
Hip fracture is a common serious injury in older adults that reduces mobility, independence, and quality of life, and can lead to premature death. Around 1.6 million cases occur globally per year, and continual increases in the number of older adults worldwide suggests that cases could reach 4.5 million by 2050. Diet can affect bone health and risk of hip fracture, with varying risks in adults on specific diets. There is some evidence that vegetarians may have poorer bone health and higher risks of fractures than meat-eaters, but prospective evidence for hip fractures is limited, and the influence of factors including diet quality and body mass index (BMI) are unclear.

The main aim of this research is to investigate risk of hip fracture in occasional meat-eaters, pescatarians, and vegetarians compared to regular meat-eaters. A secondary aim is to determine if risk of hip fracture in these diet groups depends on age, sex, diet quality, body mass index, and diet-gene interactions. Thirdly, we will explore the role of potential factors underpinning any risk differences, such as BMI, bone mineral density, and intake of nutrients that are mostly found in animal-sourced foods. The purpose of this study is to better understand hip fracture risk in vegetarian UK adults. The proposed project will use existing diet and lifestyle data from the UK Biobank resource, and hospital records of hip fractures.

DETAILED DESCRIPTION:
Background:

Hip fracture is an increasingly prevalent health problem in the UK and worldwide that increases morbidity and mortality. Previous epidemiological evidence suggests that compared to meat-eaters, people following plant-based diets have lower bone mineral density (BMD) and a higher risk of fractures. Emerging evidence suggests a higher risk of hip fracture in vegetarian women, but prospective evidence of hip fracture risk in these diet groups is scarce and limited, particularly in men. Risk differences between diet groups are plausible in men and women, for example due to bone or muscle-related nutrient deficiencies or low BMI in vegetarians, but underlying mechanisms explaining potential risk differences require further investigation.

This study aims to investigate risk of hip fracture in occasional meat-eaters, pescatarians, and vegetarians compared to regular meat-eaters in the UK Biobank cohort. A secondary aim is to determine the role of potential modifying factors on associations between each diet group and hip fracture risk, including diet quality (determined by adherence to the Alternative Healthy Eating Index, AHEI), age, sex, and BMI, as well as investigating interactions between diet groups and genotypes on BMD and hip fracture risk. Thirdly, we aim to determine the role of potential mediating factors on any observed associations, including BMI, BMD, and intake of dietary nutrients abundant in animal products.

Research plan and methods:

The investigators will utilise dietary and lifestyle data from the UK Biobank cohort, which recruited over 500,000 adults between 2006-2010, and linked hospital records of UK Biobank participants to identify hip fracture cases.

A Cox regression model will be applied to investigate risk of hip fracture in each diet group compared to regular meat-eaters, and will be adjusted for relevant confounders. The roles of age, sex, AHEI score, BMI, and diet-gene interactions as potential effect modifiers will be explored by adding each variable to Cox regression models as interaction terms. Causal mediation analysis will be used to determine the role of potential mediators.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Ages 40 to 70 years at time of recruitment
* Able to provide informed consent

Exclusion Criteria:

* Unable to link dietary and lifestyle data with hospital episode statistics
* Had a hip fracture or osteoporosis before or no the date of recruitment
* Withdrew consent during the study period
* Genetic sex differs to reported sex
* Outlier diet or anthropometric data (energy intake <500 or >5000 kcal/day or body mass index <10 or >60 kg/m2

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Information on the UK Biobank cohort profile is available here: https://www.ukbiobank.ac.uk/
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Hip fracture incidence (first) | Age when the completed questionnaire was returned (2006-2010) until age at event, death, or end of study period (2021).
  First incidence of hip fracture, identified from all relevant ICD diagnosis codes and treatment codes identified through linked HES data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD from UK Biobank is available to genuine researchers on application (https://www.ukbiobank.ac.uk/enable-your-research/apply-for-access).

REFERENCES:
- [Result] Webster J, Greenwood DC, Cade JE. Risk of hip fracture in meat-eaters, pescatarians, and vegetarians: a prospective cohort study of 413,914 UK Biobank participants. BMC Med. 2023 Jul 27;21(1):278. doi: 10.1186/s12916-023-02993-6. PMID 37501206

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT05554549/SAP_000.pdf